CLINICAL TRIAL: NCT01407445
Title: Study of the Effects of Tribulus Terrestris on Sexuality in Postmenopausal Women
Brief Title: Effects of Tribulus Terrestris on Sexual Function in Post-menopausal Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Sonia Maria Rolim Rosa Lima, Study of the Effects of Tribulus Terrestris on Sexuality in Postmenopausal Women, Faculdade de Ciências Médicas da Santa Casa de São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Fcmscsp-tribulus; terrestris (Other: CEP-008/2009)
Record Dates: First submitted 2011-08-01; First posted 2011-08-02 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Sexual Functions and Problems in the Adult
Keywords: Menopause; Sexual dysfunction; Tribulus; Sexuality; Phytotherapeutic Drugs
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Sexuality | interventions — Tribulus extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): 1 tablet of placebo/ oral/ 3 times a day for three months
  Interventions: Drug: Placebo
- Tribulus terrestris (Active Comparator): 1 tablet of 250mg/ oral/ 3 times a day for three months
  Interventions: Drug: Tribulus terrestris

INTERVENTIONS:
Drug: Placebo — 1 tablet/ oral/ 3 times a day for 90 days
  Other Names: lot 168159
  Arms: Placebo
Drug: Tribulus terrestris — 1 tablet of 250mg/ oral/ 3 times a day for 90 days
  Other Names: lot 168059
  Arms: Tribulus terrestris

SUMMARY:
Objective: To study the effects of Tribulus terrestris on sexuality in postmenopausal women.

DETAILED DESCRIPTION:
Sexuality is an integral part of every personality, influence thoughts, feelings, actions, integrations, and therefore the physical and mental health. It is estimated that 43% of women have at least one complaint of sexual problem. Disorders of desire and arousal are among the most common problems found in gynecologic practice. Medicinal plants have been used for therapeutic purposes for thousands of years, and aphrodisiac properties described in several plants. Tribulus terrestris is a plant indigenous to India, recommended in the treatment of infertility, low libido and impotence, and its main active ingredient protodioscin (PTN).

ELIGIBILITY:
Inclusion Criteria:

* Women past menopause, with full autonomy, at least one year of amenorrhea and FSH> 30 mIU / mL.
* Sexually active
* Partner is stable and without sexual difficulties
* Carrier sexual abuse (desire, arousal, orgasm and dyspareunia)

Exclusion Criteria:

* Women on hormone therapy within the preceding 12 months
* Women without sexual activity
* With diabetes mellitus
* Patients with cognitive impairment
* Patients with hormone-dependent tumor
* History of psychiatric illness
* Patients with liver disease
* Patients with kidney disease
* Users of drugs with proven to decrease sexual desire
* Cardivascular disease, renal disease.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Sexual function in post-menopausal women | 90 days
  Based the questionnaires Golombok-Rust Inventory of Sexual Satisfaction (GRISS) and Sexual Quotient - female version (SQF).

SECONDARY OUTCOMES:
Female Intervention Efficacy Index (FIEI) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Sonia lima, PhD, Principal Investigator — Faculdade de Ciências Médicas da Santa Casa de São Paulo
Locations (1):
- Santa Casa of Sao Paulo Medical School, São Paulo, São Paulo, Brazil